CLINICAL TRIAL: NCT03145493
Title: (L'Effet Des Drains Aspiratifs en Arthroplastie du Genou Avec l'Utilisation de l'Acide Tranexamique)
Brief Title: Effect of Suction Drains in Total Knee Arthroplasty With Tranexamic Acid
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CE 14.150
Record Dates: First submitted 2017-03-03; First posted 2017-05-09 (Actual); Last update posted 2020-07-17 (Actual); Status verified 2019-02

CONDITIONS: Arthroplasty, Replacement, Knee
Keywords: Drainage, Suction; tranexamic acid
MeSH Terms: interventions — Drainage

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usage of suction drains (Experimental): Usage of suction drains
  Interventions: Device: drainage
- No usage of suction drains (No Intervention): No usage of suction drains

INTERVENTIONS:
Device: drainage — Administration of IV tranexamic acid at the moment of anesthetic induction (1g) and at tourniquet release (1g), installing a suction drain
  Arms: Usage of suction drains

SUMMARY:
Problem Suction drains during TKA present certain costs to the health system and requires additional nursing care. There is no clear evidence that supports their use, and no studies so far have compared blood loss in patients with or without drains when TA is administered during TKA.

Hypothesis During total knee arthroplasty, the postoperative blood loss, measured by hemoglobin level, will be lower when no drains are used.

Method

* Randomized controlled trial
* Monocentric, 3 surgeons
* Randomisation by sealed envelopes

DETAILED DESCRIPTION:
During total knee arthroplasty, the postoperative blood loss, measured by hemoglobin level, will be lower when no drains are used.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral primary total knee arthroplasty

Exclusion Criteria:

* TKA revision
* Bilateral TKA
* Patients that refuse transfusions
* Contraindication to tranexamic acid use: allergy, thromboembolic history
* Coagulopathy
* Kidney failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2014-10-03 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
Hb variation | 3 days after surgey
  Difference between Hb levels measured in pre-op and on postoperatively day 3.

SECONDARY OUTCOMES:
Number of blood transfusions | from admission till 2 months after surgery
  Number of blood transfusions
Cost of blood transfusions | from admission till 2 months after surgery
  Cost of blood transfusions
Cost of suction drains | from admission till 2 months after surgery
  Cost of suction drains
Range of motion of knee | preoperative visit , at the end of surgery, and on post-op day 3
  Range of motion of knee
Length of hospital stay | from admission till 2 months after surgery
  Length of hospital stay
additional surgery | from admission till 2 months after surgery
  possible causes for reoperation: hematoma drainage, infection, knee mobilization
Clinical results | from admission till 2 months after surgery
  Major complications
KOOS score | At preoperative visit and post-operative visit of six weeks after surgery
  Knee Injury and Osteoarthritis Outcome Score (KOOS); Scores are transformed to a 0-100 scale, 0: extreme knee problems, 100: no knee problems
SF-12 score | At preoperative visit and post-operative visit of six weeks after surgery
  SF-12® Health Survey (SF-12); Physical and Mental Health Composite Scores (PCS & MCS) ; Minimum value: 0 (lowest level of health), Maximum value: 100 (highest level of health)

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric Lavoie, MD MSc FRCSC, Principal Investigator — CHUM
Locations (1):
- Centre Hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec, Canada